CLINICAL TRIAL: NCT05614492
Title: Development and Evaluation of a PrEP Decision Aid for Women Seeking Domestic Violence Services in Baltimore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH127986-01 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HIV; Violence, Gender-Based; Pre-Exposure Prophylaxis
Keywords: HIV Prevention; Tenofovir
MeSH Terms: interventions — SDM

STUDY DESIGN:
Intervention Model Description: Parallel: Participants will be assigned to one of three groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual Arm (IDM) (Experimental): Self-administration of the intervention
  Interventions: Behavioral: Individual PrEP Decision Aid
- Shared Arm (SDM) (Experimental): Advocate-administration of the intervention
  Interventions: Behavioral: Shared PrEP Decision Aid
- Control Arm (Time and Attention Matched Control) (Active Comparator): Self-administration of standard PrEP information from Centers for Disease Control (CDC).
  Interventions: Behavioral: CDC PrEP Video

INTERVENTIONS:
Behavioral: Individual PrEP Decision Aid — Participant engages with the decision support tool designed to optimize PrEP uptake among Black cisgender women who have experienced IPV independently. They also enter data independently.
  Other Names: IDM
  Arms: Individual Arm (IDM)
Behavioral: CDC PrEP Video — A video from the Centers for Disease Control and Prevention that provides basic, general information on PrEP
  Other Names: Control
  Arms: Control Arm (Time and Attention Matched Control)
Behavioral: Shared PrEP Decision Aid — Domestic violence service advocate (DVA) engages with the decision support tool designed to optimize PrEP uptake among Black cisgender women who have experienced IPV with the participant and enters data
  Other Names: SDM
  Arms: Shared Arm (SDM)

SUMMARY:
This study is designed to develop and test an individual decision aid for pre-exposure prophylaxis (PrEP) tailored to Black women who have been exposed to intimate partner violence and are working with a domestic violence service provider. three different ways of delivering the tailored decision aid are being tested: 1) as an individual tool; or 2) as a shared decision-making tool with a domestic violence advocate; as compared to generalized information. The goal of decision aid will be to address key cultural and structural factors affecting these women and can help them gain PrEP awareness and access.

DETAILED DESCRIPTION:
Intimate partner violence (IPV)-exposed Black women are often forced to choose between relationship safety and HIV prevention; thus, trauma-, gender-, culturally-responsive HIV prevention interventions are needed for this key priority population. Pre-exposure prophylaxis (PrEP) may be a viable partner-independent option for IPV-exposed Black women, but no study has identified an evidence-based strategy to promote and increase PrEP uptake among this population, specifically IPV-exposed Black women in the South. Guided by the Consolidated Framework for Implementation Research (CFIR), the proposed research aims to adapt, implement and evaluate self- and advocate-administered versions of a PrEP decision aid in a domestic violence agency in Baltimore in order to increase PrEP uptake among Black women in Ending the HIV Epidemic (EtHE) priority areas, address trauma as a barrier to PrEP uptake, and ultimately combat racial disparities in women's HIV cases.

Therefore, this Type II hybrid effectiveness-implementation study seeks to adapt an existing PrEP decision aid to IPV-exposed Black women seeking domestic violence (DV) services in Baltimore, an EtHE priority state. Self- and advocate-administered versions of the PrEP decision aid will be implemented and the aid will be evaluated using a three-arm randomized trial. The Consolidated Framework for Implementation Research (CFIR) will guide this research. A formative evaluation using qualitative interviews with IPV-exposed Black women (N=10) and DV advocates (N=20) was conducted to adapt the PrEP decision aid. Next, the decision aid will be implemented in a DV agency and 90 IPV-exposed Black women will be randomized to either the self- or advocate-administered versions of the aid, or the control intervention, in order to compare feasibility, acceptability and preliminary effectiveness with baseline, 1-, 3-, and 6-month surveys. Focus groups with DV advocates and participants will assess for implementation process outcomes. This study will: provide support for a PrEP decision aid that addresses HIV prevention for IPV-exposed Black women; use implementation science to increase PrEP uptake; include DV agencies in intervention development and implementation; and improve understanding of PrEP scale-up by addressing implementation factors in settings that serve IPV-exposed Black women.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* self-identification as cisgender female
* IPV-exposed (i.e., at least one physical, sexual, or psychological IPV victimization experience by a male partner) in the past 12 months
* self-reported HIV negative
* English- and/or Spanish-speaking
* self-identify as Black or African American

Exclusion Criteria:

* Currently using PrEP
* Unable to provide consent
* Participated in formative research for this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in HIV Risk Perception | Baseline and post intervention, up to 2 minutes
  8-item Perceived Risk of HIV scale repeated at the beginning and end of engagement with the decision aid, with responses measured on a 5- point Likert scale, which has been shown to be more robust than a single-item screening question for HIV risk perception. Specifically, responders will specify their level of agreement to the question in five points: (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree.
Change in Decisional preference for PrEP | Baseline and post intervention, up to 2 minutes
  Single item screening question: "How interested are you in starting PrEP now?" repeated at the beginning and end of engagement with the decision aid, with responses measured on a 5- point Likert scale, with responders specify their level of agreement to the question in five points: (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree.

SECONDARY OUTCOMES:
Change in PrEP Uptake | Month 1, Month 3, Month 6
  defined as having filled a PrEP prescription (by a composite of self-report and pharmacy refill data) and coded as a binary variable.

OTHER OUTCOMES:
Change in Feelings of Decisional conflict | Baseline, Month 1, Month 3, Month 6
  Validated measure of decision uncertainty and perceived effective decision making (i.e. about starting PrEP), specifically the healthcare consumers' decision uncertainty, the factors contributing to the uncertainty, and health-care consumers' perceived effective decision making. Utilizes a 5-point Likert scale where responders specify their level of agreement to the questions in five points: (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree.
Process Outcomes | Month 6
  A qualitative measure of: 1) feasibility of implementing the decision aid; 2) barriers and facilitators to decision aid implementation; 3) experiences conducting the decision aid or perceptions of women's experiences using decision aid; and 4) fidelity to implementation. Data collected through focus group meeting transcripts and analyzed using computer-assisted qualitative data analysis software.
Urine tenofovir levels | Month 3
  As an exploratory measure, urine Tenofovir (TFV) testing will be conducted on a sub-sample of 10 women (randomized to any arm) who start PrEP during the course of the study. Measured with a point of care lateral flow assay test with a sample collected at the Month 3 visit post-randomization to allow women sufficient time to initiate PrEP after receiving the decision aid.
Change in Feelings of Decision regret | Baseline, Month 1, Month 3, Month 6
  5-item validated instrument of personal perceptions after a healthcare decision is made (i.e. starting or not starting PrEP), with responders specify their level of agreement to the questions in five points: (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Tiara Willie, PhD, MA, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Springboard Community Services - Baltimore City Office, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No